CLINICAL TRIAL: NCT04158986
Title: Post-discharge Nurse-driven Intervention Program for Patients With Decompensated Liver Cirrhosis
Brief Title: Nurse Assisted Post-discharge Intervention in Decompensated Cirrhosis
Acronym: NurseAID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Malene Barfod O'Connell, RN, PhD student, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Splcirr2019
Record Dates: First submitted 2019-10-23; First posted 2019-11-12 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Masking Description: Allocation is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard treatment (No Intervention): Receives standard post-discharge care with planned follow-up in the clinic for liver failure or ambulatory.
- Nurse-driven post-discharge intervention (Experimental): Participates in a nurse-driven post-discharge intervention program.
  Interventions: Behavioral: Nurse-driven post-discharge intervention

INTERVENTIONS:
Behavioral: Nurse-driven post-discharge intervention — Home visits based on the concepts of Family Nursing:
  The participants will receive three home visits by a nurse who is trained in the Family Nursing principles during the first 12 weeks after discharge.
  The home visits will comprise of:
  * Filling in the Chronic Liver Disease Questionnaire.
  * Therapeutic conversations including drawing and review of genogram and eco-map.
  * Information about- and help to initiate contact to relevant municipal offers.
  * Evidence-based information based on the patient's current problems or symptoms, base-line knowledge and receptiveness.
  Follow-up telephone calls:
  • After the first 12 weeks participants will be followed-up by telephone monthly during the following 12 weeks.
  Pamphlet:
  • All participants will receive a pamphlet with brief information regarding preventive measures and early signs of decompensation as well as relevant contact details. The pamphlet will be handed out before discharge
  Arms: Nurse-driven post-discharge intervention

SUMMARY:
In a randomized controlled trial, the effects of a nurse-driven post-discharge intervention for patients with liver cirrhosis compared with standard follow-up will be investigated.

DETAILED DESCRIPTION:
Since 1970 the mortality from cirrhosis has increased with 26.7 %, with a 50% mortality rate within 2 years of diagnosis. Grave complications result in functional impairment and reduced quality of life. 20-37 % of patients with liver cirrhosis are readmitted less than 30 days after a hospitalization for decompensation. These patients have a higher 90-day mortality rate than those who avoid readmission. Re-admissions have great personal-, societal- and economic consequences.

In a randomized controlled trial, the effects of a nurse-driven post-discharge intervention for patients with liver cirrhosis, compared with standard follow-up will be investigated.

The intervention, based on concepts from Family Nursing, will comprise three home-visits within eight weeks after discharge including therapeutic conversations focusing on strengthening participants' family relationships and social networks, disease education and help to initiate contact to municipal offers. After 12 weeks the participants will be followed-up by telephone.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with liver cirrhosis and one or more complications hereto during admission to the Gastro Unit, AHH. Complications include, but are not limited to: hepatic encephalopathy, infection, ascites, edema, kidney failure, upper or lower GI bleeding.
* Patients must read and understand Danish.
* Adults >18 years.

Exclusion Criteria:

* When the diagnosis of liver cirrhosis is questioned with reasonable doubt or the diagnosis of liver cirrhosis is disproved by histology or relevant imaging.
* Patients with comorbidity as the primary diagnosis and where an independent rehabilitation or post-discharge program is offered, for example hip fracture, chronic obstructive pulmonary disease etc.
* Patients diagnosed with an active and invasive malignant disease.
* Residency outside the catchment area of Amager Hvidovre Hospital.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-10-13 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Time from discharge to first readmission. | Time from discharge to first readmission during all readmissions due to liver cirrhosis in the 6 month trial time.
  Time from discharge to first readmission.
Number of readmissions | Number of readmissions within 2 years.
  Number of readmissions within 2 years
Duration of readmissions | Duration of readmissions due to liver cirrhosis in the 6 month trial time.
  Duration of readmissions due to liver cirrhosis

SECONDARY OUTCOMES:
Health related quality of life before and after intervention | The change in health related quality of life before and after intervention (6 months trial time).
  Measured by the Chronic Liver Disease Questionnaire (CLDQ), which comprises 29 questions split into six domains. Domain scores and an overall score are presented on a 1-7 scale. Higher scores represents better HRQOL.
Self-perceived health before and after intervention | The change in self-perceived health before and after intervention (6 months trial time).
  Measured by SF-12v2® Health Survey Acute, Denmark (Danish), which comprises 12 questions split into seven domains. Higher scores represents worse self-perceived health.
Functional disability in work-, social-, and family life before and after intervention | The change in functional disability in work-, social-, and family life before and after intervention (6 months trial time)
  Measured by the Sheehan Disability Scale (SDS), which comprises three questions with scales from 0-10. Higher scores represents worse functional ability.
Mortality | The mortality rate after 6 months, 12 months and 2 years
  Mortality after 6 months, 12 months and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Malene Barfod O'Connell, RN, MScPH, Principal Investigator — Amager Hvidovre Hospital
Locations (1):
- Copenhagen University Hospital, Amager Hvidovre, Copenhagen, Hvidovre, Denmark

REFERENCES:
- [Derived] Barfod O'Connell M, Brodsgaard A, Matthe M, Hobolth L, Wullum L, Bendtsen F, Kimer N. A randomized controlled trial of a postdischarge nursing intervention for patients with decompensated cirrhosis. Hepatol Commun. 2024 Apr 26;8(5):e0418. doi: 10.1097/HC9.0000000000000418. eCollection 2024 May 1. PMID 38668732